CLINICAL TRIAL: NCT02510378
Title: Short Course Radiotherapy Combined With Chemotherapy in Stage IV Rectal Cancer With Resectable Liver Metastases
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Hua Ren, Attending physician, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CH-GI-072
Record Dates: First submitted 2015-07-12; First posted 2015-07-29 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-07

CONDITIONS: Stage IV Rectal Cancer, Liver Metastasis, Resectable
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Short course radiotherapy (Experimental): Patients with rectal cancer and resectable liver metastases receive 25 Gy in 5 fractions of 5 Gy over 5 days to the pelvis and XELOX consolidating chemotherapy (with or without target therapy) al least 4 cycles after 2 weeks.
  After evaluation, patients with resectable rectal cancer and liver metastasis will undergo surgery. Those patients with unresectable lesions will receive chemotherapy.
  Interventions: Radiation: Short course radiotherapy

INTERVENTIONS:
Radiation: Short course radiotherapy — Patients with rectal cancer and resectable liver metastases receive 25 Gy in 5 fractions of 5 Gy over 5 days to the pelvis and XELOX consolidating chemotherapy (with or without target therapy) al least 4 cycles after 2 weeks.
  After evaluation, patients with resectable rectal cancer and liver metastasis will undergo surgery. Those patients with unresectable lesions will receive chemotherapy.

SUMMARY:
Patients with rectal cancer and resectable liver metastases receive short course radiotherapy(5Gy/f x 5f) to the pelvis and XELOX consolidating chemotherapy al least 4 cycles after 2 weeks.

DETAILED DESCRIPTION:
Patients with rectal cancer and resectable liver metastases receive 25 Gy in 5 fractions of 5 Gy over 5 days to the pelvis and XELOX consolidating chemotherapy (with or without target therapy) al least 4 cycles after 2 weeks.

After evaluation, patients with resectable rectal cancer and liver metastasis will undergo surgery. Those patients with unresectable lesions will receive chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed primary carcinoma of the rectum (Lower border of tumour ≤ 10 cm from anal verge) locally advanced stage in primary site of rectum resectable synchronous liver metastases. The decision of resectable liver metastases will be made at multidisciplinary clinical meetings.

Exclusion Criteria:

* Obstruction of the gastrointestinal tract Previously constructed stoma prior radiotherapy of the pelvis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2014-01; Primary Completion 2020-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
percentage of patients undergo R0 surgery during the follow-up | 3 months

SECONDARY OUTCOMES:
The rate of early toxicity of radiotherapy according to the NCI Common Toxicity Criteria for Adverse Effects (version 3.0) | 3 months

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Dept of Radiation oncology, Cancer Hospital , Chinese Academy of Medical Science, Beijing, Beijing Municipality
  - Cancer Hospital, CAMS, Beijing